CLINICAL TRIAL: NCT04644003
Title: A Phase 1b, Double-Blind, Placebo-Controlled, First-in-Human Study to Evaluate Safety, Tolerability and Pharmacokinetics of a Two-Week Oral Treatment With STP1 in a Subgroup of Patients With Autism Spectrum Disorder
Brief Title: Safety, Tolerability and Pharmacokinetics Study of STP1 in a Subgroup of Patients With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stalicla SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STP1-C004
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- STP1 Low Dose (Experimental): 1 capsule and 1 tablet per intake
  Interventions: Drug: STP1
- STP1 High Dose (Experimental): 1 capsule and 1 tablet per intake
  Interventions: Drug: STP1
- Placebo (Placebo Comparator): 1 placebo capsule and 1 placebo tablet per intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STP1 — STP1 is a combination of two drugs, a phosphodiesterase (PDE) inhibitor and an NKCC1 inhibitor
  Arms: STP1 High Dose; STP1 Low Dose
Drug: Placebo — Placebo medication (capsule and tablet) identical in appearance to active medication
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate safety and tolerability in a subgroup of patients with Autism Spectrum Disorder (ASD). In addition, Pharmacokinetics and Pharmacodynamics, as well as efficacy of STP1 are being explored.

DETAILED DESCRIPTION:
After obtaining written informed consent, those patients who are deemed eligible for the study, will be randomized on Day 1, in a double-blinded manner, in a 3:1ratio to receive either oral STP1 (twice daily) or placebo (twice daily). The total study duration is 6 weeks, including a screening phase of up to 2 weeks, a treatment phase of 2 weeks and a post-treatment follow-up phase of 2 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female individuals, between 18 and 40 years, diagnosed of ASD.
2. Patients will be assessed for specific developmental anthropometric & anatomical criteria as well as personal and family medical history as assessed by the ASD-Phen1 semi structured interview form.
3. Patients must have a parent or reliable caregiver who can provide information about the pre-natal period and early developmental period, as required by the protocol.
4. Patient and/or parent or legal guardian willing and consenting to participate.
5. Patients with ASD and comorbid seizure disorder should be seizure-free for at least 6 months prior to screening.
6. Before enrolling in the study, subjects must agree to use double-barrier birth control methods if they engage in intercourse.

Key Exclusion Criteria:

1. Patients with an identified genetic cause of ASD in their medical record will be excluded from the study.
2. History of traumatic head injury, cerebrovascular disorder, congestive heart failure, hepatic or renal disease.
3. Thrombocytopenia.
4. Type 1 Diabetes Mellitus or uncontrolled type 2 Diabetes Mellitus, or latent autoimmune diabetes of the adult.
5. A significant risk for suicidal behavior.
6. Initiation of, or a major change in psychological / behavioral intervention within 4 weeks prior to randomization.
7. Patient with any active infection.
8. Systolic blood pressure (SBP) <80 mmHg or diastolic blood pressure (DBP) <40 mmHg or a drop in SBP of ≥20 mm Hg, or in DBP of ≥10 mm Hg, during the orthostatic recordings.
9. Clinically relevant electrocardiogram (ECG) abnormalities.
10. Clinically significant abnormal laboratory test.
11. Active clinically significant disease.
12. History of malignancy.
13. Pregnant (confirmed by laboratory testing) or lactating female patient.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Erickson CA, Perez-Cano L, Pedapati EV, Painbeni E, Bonfils G, Schmitt LM, Sachs H, Nelson M, De Stefano L, Westerkamp G, de Souza ALS, Pohl O, Laufer O, Issachar G, Blaettler T, Hyvelin JM, Durham LA. Safety, Tolerability, and EEG-Based Target Engagement of STP1 (PDE3,4 Inhibitor and NKCC1 Antagonist) in a Randomized Clinical Trial in a Subgroup of Patients with ASD. Biomedicines. 2024 Jun 27;12(7):1430. doi: 10.3390/biomedicines12071430. PMID 39062003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population is defined as ASD-Phen1 based on STALICLA criteria. The number of patients enrolled were 12 subjects with 6 subjects receiving STP1-Low Dose, 3 subjects receiving STP1-High Dose, and 3 subjects receiving placebo. All 12 subjects (100.0%) completed treatment with 0 screen failures.
Pre-assignment Details: Of 12 enrolled participants, 12 met inclusion criteria and were randomized to treatment.
Groups:
- STP1 Low Dose; STP1 High Dose: 1 capsule and 1 tablet per intake
  STP1: STP1 is a combination of two drugs, a PDE inhibitor and an NKCC1 inhibitor
Period: Overall Study
Arm/Group | STP1 Low Dose | STP1 High Dose | Placebo
Started | 6 | 3 | 3
Completed | 6 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STP1 Low Dose | STP1 High Dose | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.67 (0.82) | 19.67 (1.53) | 19.67 (2.89) | 19.17 (1.59)
Age, Continuous [Median (Full Range); unit: years] | 18.50 [18.0 to 20.0] | 20.00 [18.0 to 21.0] | 18.00 [18.0 to 23.0] | 18.50 [18.0 to 23.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 5 | 2 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 5 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated by dividing the participant's weight in kilograms by the height in metres squared.
  kg/m^2 | 36.80 (5.02) | 37.07 (6.89) | 25.17 (5.84) | 33.96 (7.38)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of Participants with Adverse Events (nature and frequency of non-serious adverse events, serious adverse events and adverse events of special interest).
Time Frame: 14 days
Population: All patients receiving at least 1 dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | STP1 Low Dose | STP1 High Dose | Placebo
Number analyzed (Participants) | 6 | 3 | 3
Participants | 6 | 3 | 3

ADVERSE EVENTS:
Time Frame: The total duration of the study for each participant was up to six weeks divided as follows: a screening phase of two weeks (from Day -14 to Day -1); a double-blind treatment phase of two weeks (from Day 1 to Day 14); and a follow-up phase of two weeks after treatment discontinuation (from Day 15 to Day 28).
Description: As per ClinicalTrials.gov definitions.
Arm/Group | STP1 Low Dose | STP1 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STP1 Low Dose (N=6) | STP1 High Dose (N=3) | Placebo (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Trichotillomania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04644003/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04644003/SAP_001.pdf